CLINICAL TRIAL: NCT07336420
Title: Treatment Patterns, Medication Usage, Effectiveness, and Safety Among US Veterans Using the Remote Electrical Neuromodulation (REN) Wearable Device for Migraine Treatment
Brief Title: Treatment Patterns Among US Veterans Using Remote Electrical Neuromodulation (REN) for Migraine Treatment
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RWE-014
Record Dates: First submitted 2026-01-11; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Migraine; PTH; Acute Treatment of Migraine
Keywords: Nerivio; Remote Electrical Beuromodulation; Medication Overuse
MeSH Terms: conditions — Migraine Disorders; Prescription Drug Overuse

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single arm, Real-World-Evidence (RWE) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nerivio treatment (Active Comparator): VA patients who were prescribed with the Nerivio REN device and treated with the device and reported baseline pain were also presented with a 2-hours post-treatment questionnaire at least twice..
  Interventions: Device: Nerivio REN device

INTERVENTIONS:
Device: Nerivio REN device — Remote electrical neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application

SUMMARY:
Among US veterans, migraine is a prevalent and disabling neurological disorder, creating a clinical need for effective treatment options.

This real-world evidence (RWE) study assessed the use, effectiveness, and safety of the REN wearable among veterans with migraine, with a primary focus on whether they need rescue medications following REN treatment. Findings from this study may help guide clinical decision-making as veterans and providers craft treatment plans that include non-pharmacologic options

DETAILED DESCRIPTION:
Migraine is a highly prevalent and disabling neurological disorder characterized by recurrent headache attacks often accompanied by nausea, sensitivity to light or sound, and functional impairmen. Affecting approximately 14% of the global population, migraine substantially reduces quality of life and interferes with daily functioning.

Within the veteran affairs (VA) population in the United States, headach disorders are particularly common, and their diagnosis has increased throughout the years. Veterans headaches mostly include both migraine and post-traumatic headache (PTH). PTH commonly develops following service-related injuries or exposures, such as service eras and traumatic brain injury (TBI), contributing their prevalence and severity. Moreover, veterans with headache disorders commonly present with multiple comorbidities, including post-traumatic stress disorder (PTSD), depression, anxiety, sleep disorders, chronic musculoskeletal pain, neck and back disorders, and TBI-related symptoms. This complex clinical profile increases disability, complicates treatment decisions, and can limit the use of certain pharmacologic therapies due to contraindications or polypharmacy.

Despite the availability of multiple therapeutic options, many patients face challenges in managing their migraine due to limited drug tolerability, contraindications, the risk of medication-overuse headache (MOH), or polypharmacy. These challenges are particularly pronounced among veterans where comorbid conditions and polypharmacy often complicate or restrict therapeutic options highlighting the need for effective, well-tolerated, non-pharmacological alternatives. Demonstrating effective pain, functional impairment and symptom relief or freedom with minimal reliance on additional medications is particularly relevant in this population. This need is supported by the adoption of non-pharmacological treatment options by the Veterans Health Administration (VHA).

Remote electrical neuromodulation (REN) is a prescribed wearable device for non-invasive, non-pharmacological treatment of migraine, indicated for acute and/or preventive treatment in patients aged 8 years and older. Many studies, including randomized controlled trials and real-world evidence have shown the efficacy and safety of the REN wearable device in treating migraine pain and associated symptoms. Given that many PTH cases present with migraine-like characteristics, VA providers may prescribe the REN wearable for PTH with migraine-like symptoms.

This real-world evidence (RWE) study assessed the use, effectiveness, and safety of the REN wearable among veterans with migraine, with a primary focus on whether they need rescue medications following REN treatment.

ELIGIBILITY:
Inclusion Criteria:

* VA patiets who were prescribed withthe Nerivio REN device
* Performed REN treatments and reported baseline and 2-hours questionnaires at least twice

Exclusion Criteria:

* None

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Rescue Medication Usage | 2 hours
  Proportion of treatments in which patients did not use additional prescribed medications within 2-hours following REN treatment

SECONDARY OUTCOMES:
Pain Relief | 2 hours
  Proportion of treatments in which there was a reduction in headache intensity from moderate or severe headache at baseline to mild or no pain 2 hours post-treatment.
Pain Freedom | 2 hours
  Proportion of treatments in which there was a reduction in headache intensity from mild or moderate or severe headache at baseline to no headache 2 hours post-treatment.
Functional Disability Relief | 2 hours
  Proportion of treatments in which there was at least one-grade improvement in functional disability level at baseline to 2 hours post-treatment.
Functional Disability Freedom | 2 hours
  Proportion of treatments in which there was a reduction in functional disability level at baseline to no functioal disability at 2 hours post-treatment.
Freedom from each migraine-associated symptom (Photophobia, Phonophobia, Nausea/Vomiting) | 2 hours
  Proportion of treatments in which there was an absence of each of the three associated symptoms 2 hours post-treatment in treatments with reported associated symptoms at baseline
Treatment intensity | 45 minutes
  Average treatment intensity across all treatments per patient and cohort
Device Safety | up to 5 years
  Rate of serious adverse events, adverse events and device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark-Inbar, PhD, Principal Investigator — Theranica
Locations (1):
- Theranica Bio-Electronics Inc, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No